CLINICAL TRIAL: NCT01515137
Title: Phase II Study of TARCEVA (Erlotinib) as Adjuvant Treatment for Locally Advanced Head and Neck Squamous Cell Carcinoma With Evaluation of Neoadjuvant Biomarker Modulation With TARCEVA vs. TARCEVA Plus Sulindac
Brief Title: Study of TARCEVA (Erlotinib) as Adjuvant Treatment for Locally Advanced Head and Neck Squamous Cell Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: OSI Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 05-045
Record Dates: First submitted 2012-01-12; First posted 2012-01-23 (Estimated); Last update posted 2023-03-28 (Actual); Status verified 2016-01

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: Head and Neck; Locally Advanced Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Erlotinib Hydrochloride; Sulindac

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm A erlotinib plus sulindac (Experimental): erlotinib (150 mg PO QD) plus sulindac (150 mg PO BID) (Arm A),
  Interventions: Drug: Erlotinib plus sulindac
- Arm B erlotinib (Experimental): erlotinib (150 mg PO QD) (Arm B)
  Interventions: Drug: Erlotinib
- Arm C (Experimental): placebo (for Erlotinib) QD (Arm C).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Erlotinib — Erlotinib (150 mg PO QD) plus sulindac (150 mg PO BID) (Arm A), Erlotinib (150 mg PO QD) (Arm B) or placebo (for Erlotinib) QD (Arm C).
  Other Names: Tarceva
  Arms: Arm B erlotinib
Drug: Erlotinib plus sulindac — Erlotinib (150 mg PO QD) plus sulindac (150 mg PO BID) (Arm A), Erlotinib (150 mg PO QD) (Arm B) or placebo (for Erlotinib) QD (Arm C).
  Other Names: Tarceva
  Arms: Arm A erlotinib plus sulindac
Drug: Placebo — Erlotinib (150 mg PO QD) plus sulindac (150 mg PO BID) (Arm A), Erlotinib (150 mg PO QD) (Arm B) or placebo (for Erlotinib) QD (Arm C).
  Other Names: Tarceva
  Arms: Arm C

SUMMARY:
This trial was originally designed and powered to compare biomarker modulation in the neo-adjuvant setting (erlotinib versus erlotinib plus sulindac versus placebo) with clinical response to erlotinib in the adjuvant setting. Since implementing the trial in late 2005, The investigators have encountered significant obstacles to implementing the adjuvant therapy phase of the trial.

* Barriers included:

  1. disease recurrence
  2. patient refusal to take the agent
  3. patient refusal to travel to Pittsburgh for clinical evaluations.

Given the institutional challenges to implement and complete the adjuvant portion, the investigators have decided to change the primary endpoint to a biomarker modulation endpoint. To achieve this goal, the investigators determined that they needed 39 paired tissue specimens (see statistical justification below).

The central hypothesis to be tested in this study is that persistent activation of parallel and/or downstream pathways contributes to tumor progression in the setting of EGFR blockade. While not all head and neck squamous cell carcinoma (HNSCC) patients will respond to EGFR targeting, the optimal strategy to identify those subjects whose tumors are sensitive to EGFR inhibition remains unknown.

The primary objective is centered around the concept of tumor biomarkers which may be modulated by EGFR and Cox-2 inhibitors and may serve as future therapeutic targets for therapy. To this end patients on this trial will be randomly assigned to one of three arms to receive either Tarceva, Tarceva plus sulindac, or a placebo in the 2 week pre-operative period. A panel of biomarkers will be obtained by biopsy prior to pre-operative therapy and again at surgery. Biomarkers will be examined for modulation in the 2-week pre-operative period, for group differences, for treatment effects and for further understanding of protein signaling pathways.

Sample size for the primary objective

Modification of Statistical Design:

The primary endpoint is the difference between pre (biopsy) and post (surgery). There are 3 hypotheses of interest: (1) placebo vs erlotinib alone, (2) placebo versus erlotinib plus sulindac, and (3) erlotinib vs erlotinib + sulindac. With a randomization in a 3:5:5 ratio, we have 88% power, alpha = .01 for an omnibus test to show between-group differences of 1 log exist. This requires 39 patients. Basically, 39 patients will provide the ability to detect a one log difference between any 2 of the 3 groups in pre-post change.

DETAILED DESCRIPTION:
Head and neck squamous cell carcinoma (HNSCC) constitutes 3 percent of all malignancies and is the sixth most common malignancy worldwide. There will be an estimated 38,000 new cases and 11,000 deaths in the United States in 2004 and approximately 500,000 cases worldwide yearly [1]. Squamous cell carcinoma accounts for at least 95 percent of all head and neck cancers. Surgical treatment remains the standard of therapy for patients with resectable HNSCC. For patients with high risk of local or distant relapse, radiation therapy (RT) alone, or in combination with chemotherapy, is given after surgery to improve loco-regional control and overall survival.

Neoadjuvant chemotherapy for patients with respectable HNSCC remains an experimental option for these patients. A two-week delay in definitive surgical resection in patients with operable HNSCC is not thought to impact the clinical outcome of these patients and in many cases may be needed to complete all of the preoperative work-up. As a result, a study design involving a two-week preoperative course of therapy in patients with operable HNSCC should not be a concern.

EGFR as a therapeutic target in HNSCC

Epidermal growth factor receptor (EGFR) is a 170-Kda transmembrane protein that is thought to be important in the proliferation and survival of cancer cells [2]. Overexpression of EGFR has been found in several malignancies, including head and neck, lung, breast, prostate, bladder, and pancreatic cancer [3-7]. In HNSCC, EGFR and its ligand TGF are overexpressed in 80-90% of tumors compared to normal mucosa; [8] the coexpression of receptor and ligand implicates an autocrine regulatory pathway in HNSCC carcinogenesis. The clinical relevance of EGFR overexpression as an independent prognostic factor in HNSCC has been well demonstrated. High tumor EGFR levels are correlated with advanced stage,[9] increased tumor size, [9] decreased survival,[10-13] increased recurrence,[10] and decreased sensitivity to radiation treatment [14]. A recent study suggests that high serum EGFR levels may even correlate with higher head and neck tumor grade [15]. The overexpression of EGFR and ligand in partially and fully transformed HNSCC tissue, its correlation with poor clinical outcome, and the aberrant function of the EGFR network in HNSCC provide compelling evidence of a relationship between EGFR and the development and progression of HNSCC, and suggest a role for EGFR as a target for cancer therapy.

EGFR has been targeted at the extracellular domain by blocking ligand binding, at the intracellular domain by inhibiting tyrosine kinase activity, and at the genetic level by targeting production of the receptor itself. EGFR-specific monoclonal antibodies interfere with ligand binding, while conjugation of an EGFR ligand or antibody to a bacterially derived toxin enables the delivery of a cytotoxic agent to the cell surface. Many of the EGFR-targeting agents are undergoing clinical evaluation in HNSCC. In general, clinical responses in HNSCC patients with advanced disease have only been observed when these agents have been combined with cytotoxic chemotherapy or radiation therapy. Clinical trials using EGFR inhibitors as adjuvant therapy for HNSCC are currently underway.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed, previously untreated HNSCC.
* Clinical stage II, III or IVA disease without distant metastasis, as defined by the American Joint Committee on Cancer Staging System, Sixth edition (See Appendix I).
* Primary tumors of the oral cavity, oropharynx, hypopharynx, or larynx will be included. Primary tumors of the sinuses, paranasal sinuses, or nasopharynx, or unknown primary tumors are NOT allowed.
* Macroscopic complete resection of the primary tumor must be planned.
* Patients will be willing to receive postoperative therapy with platinum and radiation if qualified based on criteria listed in treatment plan.
* Age 18 years.
* ECOG performance status 0-1 (See Appendix II).
* Adequate hematologic, renal and hepatic function, as defined by:

  * Absolute neutrophil count (ANC) greater than 1,500/ul, platelets greater than 100,000/ul.
  * Creatinine less than 1.5 x institutional upper limit of normal (ULN).
  * Bilirubin less than 1.5 x ULN, AST or ALT 2.5 x ULN.
* Have signed written informed consent.

Exclusion Criteria:

* Subjects who fail to meet the above criteria.
* Pregnancy or breastfeeding. Women of childbearing potential (WOCBP) must practice acceptable methods of birth control to prevent pregnancy.
* Subjects with a ECOG performance status of 2 or worse.
* Evidence of distant metastasis.
* Any other malignancy active within 5 years except for non-melanoma skin cancer or carcinoma in situ of the cervix, DCIS or LCIS of the breast.
* Prior history of HNSCC.
* Prior therapy targeting the EGFR pathway.
* Known severe hypersensitivity to sulindac or other non-steroidal anti-inflammatory drugs (NSAIDs), including aspirin.
* Any unresolved chronic toxicity greater than grade 2 from previous anticancer therapy (except alopecia), according to Common Terminology Criteria for Adverse Events v3.0 (CTCAE).
* Incomplete healing from previous major surgery.
* Acute hepatitis, known HIV, or active uncontrolled infection.
* History of uncontrolled cardiac disease; i.e., uncontrolled hypertension, unstable angina, myocardial infarction within prior 6 months, untreated known coronary artery disease, uncontrolled congestive heart failure, and cardiomyopathy with decreased ejection fraction.
* Any preexisting active interstitial lung disease (patients with chronic stable radiographic changes who are asymptomatic are NOT excluded).
* Treatment with anticoagulants, except when used to maintain the patency of a central venous line.
* Uncontrolled peptic or gastric ulcer disease, or gastrointestinal bleeding within prior 6 months.
* Active alcohol abuse or other illness that carries a likelihood of inability to comply with study treatment and follow-up.
* Treatment with a non-approved or investigational drug within 30 days prior to Day 1 of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2005-11; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Phase II Study of TARCEVA (Erlotinib) as Adjuvant Treatment for Locally Advanced Head and Neck Squamous Cell Carcinoma with Evaluation of Neoadjuvant Biomarker Modulation with TARCEVA vs. TARCEVA Plus Sulindac | 10 years
  Primary objective centered around concept of tumor biomarkers which may be modulated by EGFR & Cox-2 inhibitors & may serve as future therapeutic targets for therapy. Patients on this trial to be randomly assigned to 1 of 3 arms in the 2 week pre-operative period. A panel of biomarkers will be obtained by biopsy prior to pre-operative therapy and again at surgery. Biomarkers will be examined for modulation in the 2-week pre-operative period, for group differences, for treatment effects and for further understanding of protein signaling pathways.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Grandis, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania, United States